CLINICAL TRIAL: NCT03180957
Title: A Multi-centre, Double Blind, Randomised, Placebo-controlled, Parallel Group, Phase II Trial to Determine the Efficacy of Intra-nodular Injection of Anti-TNF to Control Disease Progression in Early Dupuytren's Disease, With a Dose Response.
Brief Title: Repurposing Anti-TNF for Treating Dupuytren's Disease
Acronym: RIDD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Department of Health, United Kingdom (Other Government); Wellcome Trust (Other); 180 Therapeutics LP (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11069; HICF-R8-433 (Other Grant/Funding Number: Health Innovation Challenge Fund); 2015-001780-40 (EudraCT Number); ISRCTN27786905 (Registry Identifier: ISRCTN); 15/SC/0259 (Other: UK Health Research Authority); CTU0028 (Other: OCTRU)
Record Dates: First submitted 2017-05-23; First posted 2017-06-08 (Actual); Results first posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2022-05

CONDITIONS: Dupuytren's Disease
Keywords: Dupuytren; adalimumab; anti TNF; phase II clinical trial; randomized controlled trial; double-blind method; Dupuytren's; Dupuytren's contracture
MeSH Terms: conditions — Dupuytren Contracture | interventions — Adalimumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: During Dose Response part of the trial the Investigator will be blinded. During the Early Disease part of the trial the Investigator will not be blinded but will not carry out any outcome assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-TNF (Experimental): adalimumab
  Interventions: Drug: Adalimumab
- Placebo (Placebo Comparator): saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Adalimumab
  Other Names: Humira
  Arms: Anti-TNF
Drug: Saline
  Arms: Placebo

SUMMARY:
Dupuytren's disease is a very common condition, affecting 4% of the general UK and US population. It causes the fingers to curl irreversibly into the palm and can be extremely disabling. The disease usually starts as a small firm lump (nodule) in the palm, and in about 40% of patients advances to form cords that pull the fingers into the palm. There is no approved treatment for the early stage of disease. Once patients have established deformities, the diseased tissue can removed by surgery or cut using less invasive techniques such as a needle or an enzyme. However, recovery following surgery usually takes several months and recurrence rates with the less invasive techniques are high.

The investigators have unravelled the cellular process that initiates and maintains the disease progress and identified tumour necrosis factor (TNF) as a new target for treatment. Based on these findings the investigators plan to test the effects of adalimumab, an anti-TNF drug which currently approved for use in patients with rheumatoid arthritis and other inflammatory conditions. The aim of the study is to find out whether treatment by injection with adalimumab directly into the diseased tissue will control the advance of early Dupuytren's disease better than a placebo injection with normal saline.

The investigators will first carry out a small trial in up to 40 patients with established disease to determine the best dose that reduces the activity of the cells responsible for the disorder (Dose Response study). In this part patients who will be having surgery to remove their diseased tissue will receive a single injection of adalimumab into the nodule in their hand about 2 weeks before surgery. The tissue that is then removed during surgery will be analysed in the investigator's laboratories to determine the effect of the drug on the tissue. Patients will be followed for 12 weeks after surgery.

In the second part of the study the investigators will assess whether the optimal dose of the drug prevents early disease advancing in 138 patients (Early Disease study). Patients who take part in the second part of the study will receive a total of 4 injections of adalimumab into the nodule in their hand at three monthly intervals. They will then be checked at 3 & 9 months after the last injection. In additional to assessing the effect of the injections on the nodule and hand function, information will also be collected to assess the cost effectiveness of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* For Part 1: Diagnosed with DD affecting the fingers resulting in flexion deformities of ≥30° at the metacarpophalangeal joint and or the proximal interphalangeal joint with impaired hand function and awaiting surgery. Or for Part 2: Participants with early disease nodules who have shown or reported progression of the disease in the previous 6 months with flexion deformities of their fingers of ≤30° at the metacarpophalangeal and/or at the proximal interphalangeal joint, i.e. total flexion deformity of up to 60°.
* The DD nodule to be treated must be distinct and identifiable.
* Female participants of child bearing potential, and male participants whose partner is of child bearing potential, must be willing to ensure that they or their partner use effective contraception throughout the treatment period and for 5 months following the last research injection. Acceptable methods of contraception include: a combination of male condom with either cap, diaphragm or sponge with spermicide (double barrier methods), injectables, the combined oral contraceptive pill (at a stable dose for at least 3 months before entering the study), an intrauterine device, vasectomised partner, or true sexual abstinence (when this is in line with the preferred and usual lifestyle of the participant).
* Participant results from safety screening tests within normal ranges within 12 weeks of enrolment, with the exception that an earlier clear chest x-ray result may be used where this is in accordance with the time frames of local standard procedures for anti-TNF screening.
* Able (in the Investigators opinion) and willing to comply with all study requirements.
* Willing to allow his or her general practitioner to be notified of participation in the study.
* Sufficient language fluency to ensure informed consent is obtained and to complete the questionnaires pertaining to hand function.

Exclusion Criteria:

* For Part 1: Participant has previously had fasciectomy, dermofasciectomy, needle fasciotomy, collagenase injection, steroid injection or radiotherapy to treat Dupuytren's disease in the digit concerned. Or for Part 2: Participant has previously had fasciectomy, dermofasciectomy, needle fasciotomy, collagenase injection, steroid injection to the digit to be treated or radiotherapy to treat Dupuytren's disease in the hand concerned.
* Female participant who is pregnant, lactating or planning pregnancy during the course of the study and for 5 months following last injection.
* Male participant who is planning a pregnancy during the course of the study and for 5 months following last injection.
* Significant renal or hepatic impairment.
* For Part 1: Scheduled elective surgery or other procedures requiring general anaesthesia during the study other than the scheduled Dupuytren's surgery. Or for Part 2: Scheduled elective surgery or other procedures requiring general anaesthesia during the study
* Participant who has ever been diagnosed with cancer, is terminally ill or is inappropriate for placebo medication
* Systemic inflammatory disorder such as rheumatoid arthritis (RA) or inflammatory bowel disease.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Participated in another research study involving an investigational medicinal product in the past 12 weeks.
* Known allergy to any anti-TNF agent.
* Have HIV or hepatitis B or C.
* Known to have an infection or history of repeated infections.
* History of Tuberculosis (TB).
* Have Multiple Sclerosis (MS) or other demyelinating disease.
* History of local injection site reactions.
* Needle phobia.
* Have moderate or severe heart failure.
* Part 1: Being treated with coumarin anticoagulants, such as warfarin.
* Have known lung fibrosis (thickening of lung tissue).
* Being treated with concomitant biologic DMARDS.
* Have received a live vaccine within the previous 4 weeks. Participants may receive concurrent vaccinations but must avoid the use of live vaccines for 12 weeks after their last injection.
* Part1: Have received parenteral steroid within the previous 6 weeks.
* Part 2: Participants at risk of Hepatitis B infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jagdeep Nanchahal, PhD FRCS, Principal Investigator — University of Oxford
Locations (3):
- The University Medical Centre, Groningen, Netherlands
- United Kingdom (2):
  - NHS Lothian, Edinburgh
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nanchahal J, Ball C, Davidson D, Williams L, Sones W, McCann FE, Cabrita M, Swettenham J, Cahoon NJ, Copsey B, Anne Francis E, Taylor PC, Black J, Barber VS, Dutton S, Feldmann M, Lamb SE. Anti-Tumour Necrosis Factor Therapy for Dupuytren's Disease: A Randomised Dose Response Proof of Concept Phase 2a Clinical Trial. EBioMedicine. 2018 Jul;33:282-288. doi: 10.1016/j.ebiom.2018.06.022. Epub 2018 Jul 6. PMID 29983350
- [Result] Nanchahal J, Ball C, Rombach I, Williams L, Kenealy N, Dakin H, O'Connor H, Davidson D, Werker P, Dutton SJ, Feldmann M, Lamb SE. Anti-tumour necrosis factor therapy for early-stage Dupuytren's disease (RIDD): a phase 2b, randomised, double-blind, placebo-controlled trial. Lancet Rheumatol. 2022 Jun;4(6):E407-E416. doi: 10.1016/S2665-9913(22)00093-5. Epub 2022 Apr 29. PMID 35949922
- [Result] Dakin H, Rombach I, Dritsaki M, Gray A, Ball C, Lamb SE, Nanchahal J. Cost-effectiveness of adalimumab for early-stage Dupuytren's disease : an economic evaluation based on a randomized controlled trial and individual-patient simulation model. Bone Jt Open. 2022 Nov;3(11):898-906. doi: 10.1302/2633-1462.311.BJO-2022-0103.R2. PMID 36378072

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anti-TNF | Placebo
Started | 70 | 70
Completed | 59 | 54
Not Completed | 11 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anti-TNF | Placebo | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 47 | 94
  >=65 years | 23 | 23 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 20 | 47
  Male | 43 | 50 | 93
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 70 | 70 | 140
alcohol consumption (Units/week) [Count of Participants; unit: Participants] — Units consumed per week with 0 being the lowest and over 35 being the highest
  Participants
    Non Drinker | 9 | 7 | 16
    up to 13 | 36 | 41 | 77
    14-35 | 23 | 20 | 43
    over 35 | 2 | 2 | 4
Current smoker [Count of Participants; unit: Participants]
  Yes | 4 | 3 | 7
  no | 66 | 67 | 133
Hand Dominance [Count of Participants; unit: Participants]
  right | 65 | 59 | 124
  left | 5 | 10 | 15
  missing | 0 | 1 | 1
Epilepsy [Count of Participants; unit: Participants]
  no | 69 | 68 | 137
  yes | 1 | 2 | 3
Liver disease [Count of Participants; unit: Participants]
  no | 70 | 70 | 140
  yes | 0 | 0 | 0
Significant exposure to occupational vibration [Count of Participants; unit: Participants]
  no | 66 | 64 | 130
  yes | 4 | 6 | 10
Previous significant trauma to affected hand [Count of Participants; unit: Participants]
  no | 57 | 56 | 113
  yes | 13 | 14 | 27
Diabetes [Count of Participants; unit: Participants]
  no | 67 | 64 | 131
  Type 1 | 0 | 1 | 1
  Type 2 | 3 | 5 | 8
Frozen Shoulder [Count of Participants; unit: Participants]
  None | 51 | 52 | 103
  Right | 6 | 6 | 12
  Left | 10 | 5 | 15
  Both Sides | 3 | 7 | 10
Ray affected by study nodule [Count of Participants; unit: Participants]
  Index | 0 | 2 | 2
  Middle | 15 | 6 | 21
  Ring | 39 | 39 | 78
  Little | 16 | 23 | 39
Affected joint [Count of Participants; unit: Participants]
  metacarpophalangeal | 54 | 60 | 114
  proximal interphalangeal | 16 | 10 | 26
Bilateral Dupytrens's disease [Count of Participants; unit: Participants]
  no | 31 | 34 | 65
  yes | 39 | 36 | 75
Treatment for Dupytren's disease in other hand [Count of Participants; unit: Participants]
  No | 53 | 56 | 109
  Yes | 17 | 14 | 31
Associated medical conditions [Count of Participants; unit: Participants]
  No | 39 | 33 | 72
  Yes | 31 | 36 | 67
  Missing | 0 | 1 | 1
Plantar Disease [Count of Participants; unit: Participants]
  No | 58 | 59 | 117
  Yes | 12 | 10 | 22
  Missing | 0 | 1 | 1
Peyronie's disease [Count of Participants; unit: Participants]
  No | 67 | 67 | 134
  Yes | 3 | 3 | 6
Garrod's Knuckle pads [Count of Participants; unit: Participants]
  No | 58 | 51 | 109
  Yes | 12 | 19 | 31
Family History (1st Degree Relatives) [Count of Participants; unit: Participants]
  No | 45 | 40 | 85
  Yes | 25 | 30 | 55

OUTCOME MEASURES:

1. Primary Outcome: Early Disease: Nodule Hardness at 12 Months
Description: Tonometry - A hardness score in arbitrary units with 0 being the lowest hardness and 100 being the greatest hardness units on a scale.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Durometer Arbitrary Units (AU)
Arm/Group | Anti-TNF | Placebo
Number analyzed (Participants) | 59 | 54
Durometer Arbitrary Units (AU) | 58.1 (11.8) | 61.2 (9.8)

2. Secondary Outcome: Early Disease: Nodule Size
Description: Measured in mm^2 where 0 is the smallest and 50 is the largest unit on a scale
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Anti-TNF | Placebo
Number analyzed (Participants) | 61 | 63
mm^2 | 21.8 (18.7) | 35.9 (28.9)

3. Secondary Outcome: Early Disease: Grip Strength
Description: Jamar meter
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Anti-TNF | Placebo
Number analyzed (Participants) | 63 | 64
kg | 34.5 (10.7) | 38.3 (11.9)

4. Secondary Outcome: Early Disease: Extension Deficit of Affected Joint
Description: Overall passive extension deficit of joint affected by treated nodule (degrees)
Time Frame: 12 months
Population: baseline were mean imputed. 12 Months: Adalimumab n=63, Saline n=65
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Anti-TNF | Placebo
Number analyzed (Participants) | 63 | 65
degrees
  Overall passive extension deficit of joint affected by treatment nodule | 3.3 (10.2) | 5.0 (12.8)
  MCP:passive extension deficit of joint affected by treated nodule: number analyzed (Participants) | 49 | 57
  MCP:passive extension deficit of joint affected by treated nodule | 0.0 (0.0) | 1.4 (5.7)
  PIP: passive extension deficit of joint affected by treated nodule: number analyzed (Participants) | 14 | 8
  PIP: passive extension deficit of joint affected by treated nodule | 14.7 (17.7) | 30.0 (20.4)

5. Secondary Outcome: Early Disease: Patient Reported Outcomes
Description: Michigan Hand Questionnaire - overall hand function with 0 as the lowest ability and 100 best possible ability units on a scale.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anti-TNF | Placebo
Number analyzed (Participants) | 64 | 66
score on a scale | 83.5 (16.1) | 78.8 (16.0)

6. Other Pre Specified Outcome: Early Disease: Analysis of Resource Use Data
Description: Patient completed questionnaire about health & social care and financial costs of Dupuytren's disease
Time Frame: 18 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from consent until 28 days after the last injection of trial, which was administered about 9 months from baseline. Therefore, adverse events were collected over approximately 10 months from baseline
Description: No related grade 3+ AEs were reported during the follow-up for this trial
Arm/Group | Anti-TNF | Placebo
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70 | 1/70
Other Adverse Events (participants affected / at risk) | 9/70 | 9/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-TNF (N=70) | Placebo (N=70)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-TNF (N=70) | Placebo (N=70)
Adverse Events (Skin and subcutaneous tissue disorders) | 6 (6) | 4 (4) — Local Itching
Adverse event (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5) — Redness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-11-21): https://cdn.clinicaltrials.gov/large-docs/57/NCT03180957/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-07): https://cdn.clinicaltrials.gov/large-docs/57/NCT03180957/SAP_001.pdf